CLINICAL TRIAL: NCT05526014
Title: The Effect of Baseline Bilateral Uterine Artery Doppler Velocimetry on Obstetric Outcomes in Hormonally Prepared Vitrified-Warmed Blastocyst Transfer Cycles: a Prospective Cohort Study
Brief Title: The Effect of Baseline Bilateral Uterine Artery Doppler Velocimetry on Obstetric Outcomes in HRT-FET Cycles
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, ŞAFAK OLGAN, Associate Professor, Akdeniz University
Other Study IDs: 49849696
Record Dates: First submitted 2022-08-31; First posted 2022-09-02 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Infertility
Keywords: Uterine artery Doppler velocimetry; Frozen - thawed embryo transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- non-pregnant: negative b-hCG results 9 days after embryo transfer.
- pregnant with obstetric complications: Patients with a positive pregnancy result who develop obstetric complications such as preeclampsia, eclampsia, fetal growth restriction, oligohydramnios, polyhydramnios, preterm birth, gestational diabetes mellitus, antenatal bleeding and etc. after the 20th gestational weeks.
- pregnant without obstetric complications: Patients who have positive pregnancy results and do not have any obstetric complications such as preeclampsia, eclampsia, fetal growth restriction, oligohydramnios, polyhydramnios, preterm birth, gestational diabetes mellitus, antenatal bleeding and etc. during pregnancy.

SUMMARY:
Researchers aim to determine how baseline (pre-conceptional) uterine perfusion characteristics affect implantation rates and obstetric complications in women who underwent high-quality blastocyst transfer.

DETAILED DESCRIPTION:
In hormonally prepared frozen embryo transfer cycles, basal bilateral uterine artery Doppler velocimetry will be performed before treatment (pre-conceptional) in each patient. Only patients who have high-quality blastocyst stage embryos will be included in the study. Since the implantation potential of the specified embryos is high, possible embryo-induced implantation failure would be minimized.

Bilateral uterine artery Doppler velocimetry will be performed during the basal ultrasonography (on the 2-5th day of menstruation). Any uterine artery notch, absent diastolic or reverse flow also will be recorded. In addition, sub-endometrial (arcuate artery) blood flows will be evaluated by Doppler ultrasonography.

For endometrial preparation, estrogen replacement will be given for approximately 12-14 days as a routine In cases with endometrial thickness ≥7mm, progesterone treatment will be started and embryo transfer will be planned on the 6th day of the treatment.

A pregnancy test will be performed 9 days after embryo transfer. Pregnant patients will be called for ultrasonography control 3 weeks later to determine fetal heartbeat. Additionally, the patients will be followed till labor and any obstetric complications will be recorded.

Uterine artery Doppler ultrasonography findings in patients with and without pregnancy will be compared. Additionally, in the group in which pregnancy was achieved, obstetric results including birth weight, small-large for gestational age, presence of hypertension, and preterm labor will be correlated with baseline (pre-conceptional) uterine artery Doppler parameters.

ELIGIBILITY:
Inclusion Criteria:

* Exogenous hormone preparation of the endometrial lining
* High embryo quality ((≥2BB) according to Alpha criteria
* Embryo transfer at the blastocyst stage

Exclusion Criteria:

* Patients whose treatments were canceled for any reason before the embryo transfer procedure
* Patients who underwent embryo transfer in the cleavage stage
* Presence of low-quality (<2BB) blastocysts
* >15% loss of viability of the embryo during embryo thawing,
* Patients with congenital uterine malformations,
* Patients in whom Doppler velocimetry cannot be performed optimally

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All patients who have artificial endometrial preparation with high-quality blastocysts between May 2022 and December 2022 will be included. All included patients will have bilateral uterine artery Doppler velocimetry on 2-5 days of their menstrual cycle by transvaginal ultrasonography.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Live Birth Rate | 9 months
  pregnancy beyond 24 weeks of gestational age.
Obstetric Complication Rates | 24th gestational weeks till delivery
  Conditions such as preeclampsia, eclampsia, fetal growth restriction, oligohydramnios, polyhydramnios, preterm birth, gestational diabetes mellitus, antenatal bleeding and etc. that develop during pregnancy

SECONDARY OUTCOMES:
Positive β-hCG results | Nine days after each embryo transfer
  Positive β-hCG results nine days after embryo transfer.

CONTACTS AND LOCATIONS:
Overall Officials: ŞAFAK OLGAN, MD, Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)